CLINICAL TRIAL: NCT00781079
Title: Promoting Recovery Using Mental Health Consumer Providers
Brief Title: Do Consumer Providers Enhance Recovery?
Acronym: PEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 06-227
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Mental Disorder
Keywords: Organization Innovation; Opinion Leaders; Schizophrenia
MeSH Terms: conditions — Mental Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Consumer Provider (Experimental): Adding a Consumer Provider to Intensive Case Management Teams (called MHICM in the VA)
  Interventions: Behavioral: Consumer Provider
- Care as Usual (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Consumer Provider — Adding a Consumer Provider to Intensive Case Management Teams (called MHICM in the VA)
  Arms: Consumer Provider

SUMMARY:
Serious mental illness (SMI) is the second most costly disorder treated in the VHA, yet clinical outcomes for these patients in public sector settings are often poor due to a combination of low quality care and severe cognitive and functional impairments evidenced by this group. While these problems are multifaceted, studies outside the VHA have shown that using "consumer providers" (CPs) can improve and augment public care. Similar to recovering addiction counselors, CPs are individuals with SMI who use their lived experiences to provide services to others with SMI. CPs can reach out to patients that are difficult to engage, assist patients with tasks of daily living, offer a variety of rehabilitation (vocational, social, residential) services, be role models and offer hope for recovery, and facilitate support groups. Randomized controlled and quasi-experimental trials, all done outside the VHA, have shown that CPs can provide services that yield at least equivalent patient outcomes with particular benefits noted on intensive case management teams. Based on these successes both the President's New Freedom Commission and the Veteran Administration's Mental Health Strategic Plan call for broader dissemination of CPs as way to make mental health services more recovery-oriented, a recent national priority. Because of these recent calls, employing mentally ill veterans has just begun, although no effort has been made to evaluate their impact inside the VA mental health system. Yet its success outside the VHA and the recent emphasis on recovery-oriented care suggests the need to test this model in the VHA.

DETAILED DESCRIPTION:
Background/Rationale Serious mental illness (SMI) is the second most costly disorder treated in the VHA, yet clinical outcomes for these patients are often poor due to a combination of low quality care and severe cognitive and functional impairments. While these problems are multifaceted, studies outside the VHA have shown that using "consumer providers" (CPs) can improve and augment care. Similar to recovering addiction counselors, CPs are individuals with SMI who use their lived experiences to provide services to others with SMI. CPs can reach out to patients that are difficult to engage, assist patients with tasks of daily living, offer a variety of rehabilitation (vocational, social, residential) services, be role models and offer hope for recovery, and facilitate support groups. Randomized controlled and quasi-experimental trials outside the VHA have shown that CPs can provide services that yield at least equivalent patient outcomes with particular benefits noted on intensive case management teams. VHA has hired about 250 CPs to date, although their impact has not been documented. Yet its success outside the VHA and the recent emphasis on recovery-oriented care suggests the need to test this model in the VHA.

Objectives To conduct a randomized controlled trial testing the impact on patient level and team level outcomes of the implementation of CP services on six mental health intensive case management (MHICM) teams in VISN-22. The specific aims were to: 1) Evaluate the acceptability, facilitators of and barriers to the inclusion of two CPs to each intervention MHICM team. 2) Evaluate the effect of including CPs on the degree to which MHICM teams services are recovery-oriented. 3) Evaluate the effect of including CPs on veterans' clinical and recovery-focused outcomes. Our hypotheses were that CPs would be feasible and acceptable, that teams would become more recovery-oriented, and that the involvement of CPs would lead to greater gains in recovery, quality of life, empowerment with regard to illness, and to a lesser extent, symptoms compared to patients on teams without CPs.

Methods This project was a "cluster randomized controlled trial" comparing 3 CP-MHICM teams (with CPs) to 3 control teams (i.e., without a CP), at MHICM sites within VISN-22. All patients on the 6 MHICM teams' caseload during each site's recruitment period were eligible. 282 MHICM patients were enrolled, 149 at the intervention sites and 133 at the control sites. Each intervention MHICM team used a strategic planning process to tailor the CP intervention to local priorities and structures, involving multiple meetings to discuss the CP's role, hiring, and incorporation of CPs into the team. The project hired the CPs, provided training, assisted in their implementation on the teams and provided ongoing supervision. The CPs worked for about 12 months.

Using a patient survey, the study assessed impacts of CPs on patient level outcomes including recovery-orientation of their team (Recovery Self-assessment scale), individual recovery (Mental Health Recovery Measure, Illness Self-Management Scale), quality of life (Quality of Life Interview), symptoms (BASIS-24), and patient activation (Patient Activation Measure). The patient level outcome assessments were conducted pre and post intervention. Final follow-up assessment rates ranged from 71- 95% at intervention sites and 80 - 88% at control sites.

We conducted site visits with all six MHICM teams using a validated, standardized protocol, rating each team's level of recovery orientation before and after the deployment of the CPs on the Recovery-Oriented Practices Index (ROPI). We conducted 23 focus groups and interviews with patients, providers and CPs at all intervention sites (about 8 per site) at the post time point to assess barriers and facilitators to CP implementation. All focus groups and interviews were recorded, transcribed, and coded using Atlas.ti.

The analyses of the patient survey data were comparisons of changes between baseline and followup scores with regression analyses of the change scores for all the outcomes mentioned above. The first analyses was whether the intervention group was significantly related to change considering only treatment group and statistically controlling for baseline score. The second was the same as the first, adding demographics (age, gender, race, living situation and education level) and site as fixed covariates. The ROPI ratings were made on a very small number of units (6 teams), therefore the results were descriptive and involved a percent change from pre to post. The focus groups and interviews were each summarized and then summarized by site. The study team discussed the results. Using the constant comparison method, salient topics were compared within and across roles and sites.

Status Completed. Major activities and accomplishments included hiring 6 CPs who together logged over 2000 clinical encounters over the funding period of the project.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a Serious Mental Illness;
* Patient must be working with a VA Intensive Case Management team

Exclusion Criteria:

* Prior exposure to intervention; Reduced capacity;
* Patient is no longer working with a VA Intensive Case Management

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Chinman, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA; Amy N. Cohen, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (7):
- United States (7):
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Chinman M, Shoai R, Cohen A. Using organizational change strategies to guide peer support technician implementation in the Veterans Administration. Psychiatr Rehabil J. 2010 Spring;33(4):269-77. doi: 10.2975/33.4.2010.269.277. PMID 20374985
- [Result] Chinman M, Salzer M, O'Brien-Mazza D. National survey on implementation of peer specialists in the VA: implications for training and facilitation. Psychiatr Rehabil J. 2012 Dec;35(6):470-3. doi: 10.1037/h0094582. PMID 23276242
- [Result] Chinman M, Oberman RS, Hanusa BH, Cohen AN, Salyers MP, Twamley EW, Young AS. A cluster randomized trial of adding peer specialists to intensive case management teams in the Veterans Health Administration. J Behav Health Serv Res. 2015 Jan;42(1):109-21. doi: 10.1007/s11414-013-9343-1. PMID 23657754
- [Result] Hamilton AB, Chinman M, Cohen AN, Oberman RS, Young AS. Implementation of consumer providers into mental health intensive case management teams. J Behav Health Serv Res. 2015 Jan;42(1):100-8. doi: 10.1007/s11414-013-9365-8. PMID 24091610
- [Result] Chinman M, George P, Dougherty RH, Daniels AS, Ghose SS, Swift A, Delphin-Rittmon ME. Peer support services for individuals with serious mental illnesses: assessing the evidence. Psychiatr Serv. 2014 Apr 1;65(4):429-41. doi: 10.1176/appi.ps.201300244. PMID 24549400
- [Result] Chinman M, Oberman RS, Hanusa BH, Cohen AN, Salyers MP, Twamley EW, Young AS. Erratum to: A Cluster Randomized Trial of Adding Peer Specialists to Intensive Case Management Teams in the Veterans Health Administration. J Behav Health Serv Res. 2015 Jan;42(1):122. doi: 10.1007/s11414-013-9377-4. No abstract available. PMID 24217992
- See also: Paper linked to the study — http://www.ncbi.nlm.nih.gov/pubmed/16645906

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Consumer Provider | Care as Usual
Started | 149 | 133
Completed | 122 | 116
Not Completed | 27 | 17

BASELINE CHARACTERISTICS:
Population: Veteran patients of MHICM teams
Groups:
- Total: Total of all reporting groups
Arm/Group | Consumer Provider | Care as Usual | Total
Number analyzed (Participants) | 149 | 133 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of enrollment
  years | 54.59 (9.19) | 51.89 (11.13) | 52.95 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 134 | 116 | 250
Race/Ethnicity, Customized [Number; unit: participants]
  African American non-Hispanic | 39 | 13 | 52
  White non hispanic | 74 | 78 | 152
  Bi racial non hispanic | 10 | 12 | 22
  African American Hispanic | 1 | 1 | 2
  White Hispanic | 18 | 21 | 39
  Unknown | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149 | 133 | 282

OUTCOME MEASURES:

1. Primary Outcome: BASIS-R
Description: The BASIS-R is a 24 item, comprehensive instrument assessing a range of psychiatric symptoms and problems. It is valid and reliable in both inpatient and outpatient settings in populations with SMI. All items have five response options ranging from 0 to 4, with higher scores indicating more problems (range in possible scores is 0 to 96).
Time Frame: immediately before the intervention (BL), and 12 months post intervention (Post).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Care as Usual: Care as usual on the case management teams
Arm/Group | Consumer Provider | Care as Usual
Number analyzed (Participants) | 122 | 116
units on a scale
  baseline | 26.15 (14.28) | 29.34 (14.24)
  Post | 24.57 (14.05) | 26.76 (15.11)
Statistical Analysis 1: Comparison: Consumer Provider vs Care as Usual; comparisons between the PS and Usual Care groups were completed with a regression testing the interaction of group (PS vs Usual Care) and time (baseline vs follow-up) for the outcome measure. The measure was analyzed with mixed effect hierarchical regressions which accounted for the nesting of site under treatment, subjects within sites, and subjects over time; Test type: Superiority or Other; p = .5, Regression, Linear — Models included site, age, race, ethnicity

2. Secondary Outcome: Mental Health Recovery Measure (MHRM)
Description: The Mental Health Recovery Measure (MHRM) is a 30-item, 5-point behaviorally-anchored self-report measure based upon recovery experiences of persons with psychiatric disabilities. The MHRM total score has good validity, correlating strongly with the Empowerment Scale and Community Living Skills Scales, yet assessing unique aspects of recovery. Range of total score is 0 to 144, with higher scores meaning better recovery.
Time Frame: immediately before the intervention (BL), and 12 months post intervention (Post).
Population: comparisons between the PS and Usual Care groups used a regression testing the interaction of group (PS vs Usual Care) and time (baseline vs follow-up) for the outcome measure. The measure was analyzed with mixed effect hierarchical regressions which accounted for the nesting of site under treatment, subjects within sites, and subjects over time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Consumer Provider | Care as Usual
Number analyzed (Participants) | 122 | 116
units on a scale
  Baseline | 85.00 (17.88) | 78.3 (18.79)
  Post | 85.66 (15.9) | 80.52 (16.54)
Statistical Analysis 1: Comparison: Consumer Provider vs Care as Usual; Test type: Superiority; p = .56, Regression, Linear; Z tests if Reg coeff are diff from 0 = -.58

3. Secondary Outcome: Patient Activation Measure
Description: The mental health version of the Patient Activation Measure (PAM) is a single 13-item scale designed to assess patient's knowledge, skill, and confidence in health self-management. Respondents endorse items (e.g., "I know what each of my prescribed medications do") on a scale from 1 ("disagree strongly") to 4 ("agree strongly"). Raw scores are converted using the established methodology for the PAM to an activation score from 0 (lowest)-100 (highest). Identifying levels of activation is based on whether an activation score falls within a previously determined range of scores. Level 1, the lowest level of activation, includes activation scores of 47 or lower; Level 2 includes scores of 47.1 to 55.1; Level 3 includes scores of 55.2 to 67.0; and Level 4 (the highest activation level) includes scores of 67.1 or above. This version has similar psychometric properties as the original 13-item PAM and correlates with related constructs in other samples of people with SMI.
Time Frame: immediately before the intervention (BL), and 12 months post intervention (Post).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Consumer Provider | Care as Usual
Number analyzed (Participants) | 122 | 116
units on a scale
  baseline | 39.31 (5.41) | 39.09 (5.37)
  post | 40.34 (5.5) | 38.76 (5.01)
Statistical Analysis 1: Comparison: Consumer Provider vs Care as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .05, Regression, Linear — Models included site, age, race, ethnicity. This is the calculated p value

4. Secondary Outcome: Recovery Self-Assessment: Person in Recovery Version
Description: Perceptions of the recovery orientation of the program were assessed with the Recovery Self-Assessment (RSA), a 36 item survey that assesses domains of recovery-orientated practice (e.g., focus on life goals, involvement of patients in their own care). The RSA has high internal consistency and is thought to represent a more recovery-oriented or recovery-supportive environment. Each item ranges from 1 to 5. The total score (all 36 items averaged together) also is reported on that scale, with higher meaning more recovery.
Time Frame: immediately before the intervention (BL), and 12 months post intervention (Post)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Consumer Provider | Care as Usual
Number analyzed (Participants) | 122 | 116
units on a scale
  Baseline | 3.86 (.53) | 3.81 (.61)
  Post | 3.93 (.61) | 3.83 (.52)
Statistical Analysis 1: Comparison: Consumer Provider vs Care as Usual; Test type: Superiority; p = .58, Regression, Linear; Z test if reg coeff is diff from 0 = .56

5. Secondary Outcome: Illness Management and Recovery Scale: Client Self-Rating
Description: The Illness Management and Recovery Scale (IMR) has 15 items (rated on 5-point behaviorally anchored scales) that assess progress toward goals, knowledge about mental illness, involvement with significant others and self-help, time in structured roles, impairment in functioning, symptom distress and coping, relapse prevention and hospitalizations, use of medications, and alcohol and drug use. A total IMR score is made of the mean of the items and has demonstrated good internal consistency, stability (test-retest after two weeks), and convergent validity, correlating with the Recovery Assessment Scale and the Colorado Symptom Index. The total score is reported on the scale of 1 to 5 with higher scores mean better recovery.
Time Frame: 12 months prior to the intervention (BL1), immediately before the intervention (BL2), and 12 months post intervention (Post).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Consumer Provider | Care as Usual
Number analyzed (Participants) | 122 | 116
units on a scale
  Baseline | 3.51 (.58) | 3.39 (.56)
  Post | 3.56 (.56) | 3.48 (.54)
Statistical Analysis 1: Comparison: Consumer Provider vs Care as Usual; Test type: Superiority; p = .87, Regression, Linear; Z test if reg coeff is diff than 0 = -.16

6. Secondary Outcome: Quality of Life Interview, Brief Version
Description: Subjective ratings of overall quality of life and the quality of social relationships, daily life, and family interactions was assessed using a combination of selected scales from the Quality of Life Instrument-Brief Version (QOLI), which been used extensively with a wide range of populations including those who are homeless, have a dual diagnosis, and are ethnic minorities. Because of low internal consistencies of subscales in our sample, a factor analysis was conducted which indicated that a larger scale that included the items from the overall quality of life, social relationships, daily life, and family interactions scales would be more reliable (all items averaged together). The score ranges from 1 to 5, with 1 meaning more quality of life.
Time Frame: immediately before the intervention (BL), and 12 months post intervention (Post).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Consumer Provider | Care as Usual
Number analyzed (Participants) | 122 | 116
units on a scale
  Baseline | 4.64 (1.04) | 4.54 (1.03)
  Post | 4.72 (1.04) | 4.71 (.9)
Statistical Analysis 1: Comparison: Consumer Provider vs Care as Usual; Test type: Superiority; p = .98, Regression, Linear; Z test if ref coeff is diff than 0 = .03

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Case as Usual: Care as usual on case management teams
Arm/Group | Consumer Provider | Case as Usual
Serious Adverse Events (participants affected / at risk) | 85/149 | 55/133
Other Adverse Events (participants affected / at risk) | 0/149 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Consumer Provider (N=149) | Case as Usual (N=133)
Death (Cardiac disorders) | 10 (10) | 3 (3)
Psychiatric (Psychiatric disorders) | 41 (105) | 23 (74)
Cardiac (Cardiac disorders) | 24 (45) | 10 (12)
other hospitalizations (General disorders) | 10 (40) | 19 (19)

LIMITATIONS AND CAVEATS:
1. cluster randomized trial - teams may have exerted influence on the findings. 2. analyses were intent-to-treat, but about half the veterans in the PS group did not receive any PS services. 3. the study involved a small number of peers (n=6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes